CLINICAL TRIAL: NCT03290989
Title: Itch and Pain Characteristics in Skin Carcinomas
Acronym: PRURITCC
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PRURITCC
Record Dates: First submitted 2017-09-14; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Skin Carcinoma; Skin Cancer; Pruritus
MeSH Terms: conditions — Skin Neoplasms; Pruritus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to have better knowledge about sensations of patients with skin carcinomas and to have data about characteristics of pain and pruritus . All patients presenting with a suspicions lesion for skin carcinomas will be included and will respond to a questionnaire. Demographics data, and histological data about skin carcinomas will be collected.

ELIGIBILITY:
Inclusion Criteria:

all patients with suspected skin carcinoma aged 18 years or more

Exclusion Criteria:

* age under 18 years,
* inability to complete the questionnaire because of cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 1 April 2015 to 31 July 2015, all patients presenting with a skin lesion suspicious for carcinoma (BCC or SCC) at the Department of Dermatology of the Military Hospital in Brest were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluate characteristics of pruritus in skin carcinomas | Day1 (when presenting at consultation with a skin lesion suspicious for carcinoma)
  Questions about characteristics
Evaluate characteristics of pruritus in skin carcinomas | Day1 (when presenting at consultation with a skin lesion suspicious for carcinoma
  Numerical visual scale (EVA)
Evaluate characteristics of pruritus in skin carcinomas | Day1 (when presenting at consultation with a skin lesion suspicious for carcinoma
  5D-itch scale
Evaluate characteristics of pain in skin carcinomas | Day1 (when presenting at consultation with a skin lesion suspicious for carcinoma
  Numerical visual pain
Evaluate characteristics of in skin carcinomas | Day1 (when presenting at consultation with a skin lesion suspicious for carcinoma
  score DN4

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France